CLINICAL TRIAL: NCT07059611
Title: Phase II Study of Neoadjuvant RP2 in Combination With Preoperative Flot for Patients With Stage II or Higher, Non-metastatic Gastroesophageal Adenocarcinoma
Brief Title: Neoadjuvant Intra-tumoral RP2 and FLOT in Gastroesophageal Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Replimune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 06225
Record Dates: First submitted 2025-07-08; First posted 2025-07-11 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Gastric Adenocarcinoma; Esophageal Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Docetaxel; pegfilgrastim; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RP2 and FLOT (Experimental)
  Interventions: Biological: RP2; Combination Product: 5-Fluorouracil; Combination Product: Leucovorin; Combination Product: Oxaliplatin; Combination Product: Docetaxel; Drug: Pegfilgrastim; Drug: Filgrastim; Procedure: Surgical Resection of Primary Tumor

INTERVENTIONS:
Biological: RP2 — Upper endoscopy with RP2 intra-tumoral injection of 1 x 10(6) plaque forming units (PFU)/mL for first intra-tumoral injection, up to 10mL of 1x107 PFU/mL of RP2 for subsequent intra-tumoral injections. Injection will occur within 4 days prior of each cycle FLOT.
Combination Product: 5-Fluorouracil — 5-Fluorouracil as part of the FLOT regimen 2,600mg/m2 intravenous infusion over 24 hours on day 1 of each 14-day cycle for 4 cycles.
Combination Product: Leucovorin — Leucovorin as part of the FLOT regimen 200mg/m2 intravenous infusion on day 1 of a 14-day cycle for 4 cycles.
Combination Product: Oxaliplatin — Oxaliplatin as part of the FLOT regimen 85mg/m2 intravenous infusion on day 1 of a 14-day cycle for 4 cycles.
Combination Product: Docetaxel — Docetaxel as part of the FLOT regimen 50mg/m2 intravenous infusion on day 1 of a 14-day cycle for 4 cycles.
Drug: Pegfilgrastim — Pegfilgrastim or Filgrastim is required on the study and should be administered per the package insert of the commercially obtained drug following each cycle of FLOT for 4 cycles.
Drug: Filgrastim — Filgrastim or Pegfilgrastim is required on the study and should be administered per the package insert of the commercially obtained drug following each cycle of FLOT for 4 cycles.
Procedure: Surgical Resection of Primary Tumor — Following 4 cycles of preoperative FLOT with RP2 injections, surgical resection of esophageal, GEJ, or gastric primary tumor per standard of care practice.

SUMMARY:
The research study is being conducted to study whether performing injections of a new treatment, called RP2, directly into stomach and esophagus tumors along with standard chemotherapy (called FLOT) is safe and whether it does a better job of killing cancer before surgery compared to chemotherapy alone.

DETAILED DESCRIPTION:
This is a single-arm, phase II study using a Simon two-stage optimal design with a 6 patient safety run-in evaluating the addition of intra-tumoral injections of RP2 to standard of care perioperative FLOT for patients with stage II or higher, non-metastatic esophageal, gastroesophageal junction (GEJ), or gastric adenocarcinoma. We hypothesize that the addition of RP2 to perioperative FLOT will be safe and will significantly improve pathologic complete response (pCR) rate compared to the historical weighted average of 12% observed with perioperative FLOT in the ESOPEC trial, MATTERHORN trial, and FLOT4 trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed and clinically staged T2 or higher or node positive, non-metastatic esophageal, gastroesophageal junction, or gastric adenocarcinoma.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1.
* Patents must be deemed a surgical candidate by a thoracic surgeon, surgical oncologist, or surgeon who is qualified to perform the appropriate surgical procedure based on patient's primary tumor site.
* Patients must have normal organ and bone marrow function, as defined below, less than or equal to 14 days prior to the initiation of study therapy:

  * Absolute neutrophil count (ANC) ≥ 1,500/microliter
  * Platelets ≥100,000/microliter
  * Total bilirubin ≤ the institutional upper limit of normal (ULN).
  * AST and ALT ≤ 2.5 times the institutional ULN
  * Serum creatinine ≤ 1.5 times the institutional ULN
  * Hemoglobin ≥ 9 g/dL

Exclusion Criteria

* Has received prior chemotherapy, radiation therapy, or immunotherapy (anti-programmed cell death protein-1 (PD-1), anti-programmed death ligand-1 (PD-L1), or anti-cytotoxic T-lymphocyte associated protein 4 (CTLA-4) for the current malignancy.
* Per the investigator, has contraindications to receiving chemotherapy with FLOT.
* Per the sub-investigator (gastroenterologist) responsible for intra-tumoral injections or the investigator, patient has contraindications to repeated upper endoscopy for intra-tumoral injections. These could include medical conditions that would, per the judgment of the sub-investigator or investigator, inappropriately increase the risk of upper endoscopy.
* Conditions in which anticoagulant therapies cannot be safely stopped in the periprocedural period or patients on warfarin with a target international normalized ratio (INR) ≥ 2.5 that cannot be temporarily reversed to INR ≤ 1.7.
* Active significant herpetic infections or prior complications of Herpes simplex virus-1 (HSV-1) infection (e.g., herpetic keratitis or encephalitis) or requires intermittent or chronic use of systemic (oral or intravenous [IV]) antivirals with known antiherpetic activity (e.g., acyclovir). Note: Patients with sporadic cold sores may be enrolled as long as no active cold sores are present at the time of first dose of study treatment.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacille Calmette-Guérin (BCG), and typhoid vaccine. Note: Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed, however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. Available COVID-19 vaccines do not contain live virus and are allowed.
* Has a condition requiring systemic treatment with corticosteroids (>10mg/day prednisone equivalents) or other immunosuppressive medications within 14 days of first study treatment administration.

  * Inhaled or topical steroids and adrenal replacement doses ≤ 10mg/day of prednisone equivalents are permitted.
* Prior organ transplantation including allogeneic stem-cell transplantation.
* Has a previous or concurrent malignancy. Exceptions include:

  * Non-melanoma skin cancer, in situ cervical cancer, superficial bladder cancer, or breast cancer in situ OR
  * Prior malignancy has been completely excised or removed and patient has been continuously disease free for > 5-years
* Has a positive test result for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection with hepatitis B or hepatitis C. Testing will be performed as part of screening on the study.

  * Patients with a known history of hepatitis B or hepatitis C that have been effectively treated (with negative HBsAg and HCV RNA) will be eligible for enrollment on this criterion.
* Has a known history of human immunodeficiency virus (HIV) with detectable viral load. HIV testing will not be performed as part of screening for the study.

  * Patients with known HIV infection with an undetectable viral load and who are on a stable highly active antiviral regimen per the investigator's assessment will eligible to enroll.
* Has a psychiatric illness, substance use, or other social conditions that, in the judgment of the investigator, would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response | Assessed after completion of neoadjuvant FLOT and intra-tumoral injections of RP2 and surgical resection. This will typically be in the range of 4-5 months from the time of enrollment.
  Pathologic complete response defined as the absence of residual invasive cancer on histologic examination of the resected esophageal, GEJ, or gastric adenocarcinoma specimen and all sampled regional lymph nodes. This will be assessed in the efficacy population who received at least three intra-tumoral injections of RP2 and underwent subsequent surgical resection.

SECONDARY OUTCOMES:
Adverse event profile | The adverse event reporting period first RP2 intratumoral injection until 30 days post-surgical resection or 56 days after the last administration of RP2 (if no resection or or consent withdrawal).
  Frequency of adverse events as categorized and graded per Common Terminology Criteria for Adverse Events (CTCAE) v5.0 in patients who received at least one dose of study treatment (Safety population).
R0 resection rate | Assessed after completion of neoadjuvant FLOT and intra-tumoral injections of RP2 and surgical resection. This will typically be in the range of 4-5 months from the time of enrollment.
  R0 resection defined as a complete resection with histologically negative margins with no macroscopic or microscopic residual tumor left behind after resection (Efficacy population).
Disease-free Survival (DFS) | Follow up for this end point may occur for up to 5 years following surgical resection, or data cutoff, whichever comes first.
  DFS defined as time from surgical resection of esophageal, GEJ or gastric cancer to death or documented disease recurrence with censoring at the time of last patient contact if lost to follow up, or at the time of data cutoff (Efficacy population).
Overall Survival (OS) | Follow up for this end point may occur for up to 5 years following surgical resection, or data cutoff, whichever comes first.
  OS defined as the time from first study treatment to death with censoring at the time of last patient contact if lost to follow up, or at the time of data cutoff (Safety population).

OTHER OUTCOMES:
Exploratory | Blood plus/minus tissue samples will be collected during the preoperative FLOT and RP2 injection, at surgical resection, and the first cycle of post-operative FLOT. These collections will occur within the first 6-8 months on the study.
  Blood and tissue samples will be collected, processed, and stored. Endpoints may include pre-/post-treatment change in circulating immune cell subsets, pre-/post-treatment change in tumor infiltrating immune cell subsets, and pre-/post-treatment change in tumor gene expression profiling. These findings will also be evaluated for association with response to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: William Chapin, MD, MSCE, Principal Investigator — Abramson Cancer Center at the University of Pennsylvania
Locations (1):
- Abramson Cancer Center at the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the clinical trial publication, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months following clinical trial publication. No end date.
Access Criteria: To achieve aims in an approved proposal. Proposals should be directed to corresponding author on the clinical trial publication.